CLINICAL TRIAL: NCT05241691
Title: Retrospective Clinical Study for the Evaluation of the Safety and Clinical Performance of the Medical Device "Guided Growth Plate System Plus" (GGPSP) for the Treatment of Bone Deformities of the Lower Limbs in Skeletally Not Mature Children.
Brief Title: Retrospective Evaluation of Guided Growth Plate System Plus's Safety and Clinical Performance for the Treatment of Lower Limbs Deformities.
Status: Completed | Type: Observational
Sponsor: Orthofix s.r.l. (Industry)
Responsible Party: Sponsor
Other Study IDs: OCI_2101
Record Dates: First submitted 2022-02-02; First posted 2022-02-16 (Actual); Results first posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Genu Varum; Genu Valgum; Joint Diseases; Knee Deformity; Ankle Deformity; Length Inequality, Leg; Discrepancy Length; Congenital; Deformity of Limb
Keywords: pediatric; 8-Plate Plus; hemiepiphysiodesis; epiphysiodesis; guided growth
MeSH Terms: conditions — Genu Varum; Genu Valgum; Joint Diseases; Leg Length Inequality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients treated with Guided Growth Plate System Plus: Pediatric patients treated with Guided Growth Plate System Plus (GGPSP) for the correction of femur and/or tibia deformities
  Interventions: Device: Guided Growth Plate System Plus

INTERVENTIONS:
Device: Guided Growth Plate System Plus — The implant is thought as one of the surgical options to perform epiphysiodesis and hemiepiphysiodesis minimally invasive, that is without recourse to a corrective osteotomy.
  Other Names: 8-Plate Plus

SUMMARY:
Orthofix is conducting this retrospective Post-market clinical follow up (PMCF) study to assess the safety and clinical performance of the Guided Growth Plate System Plus (GGPSP) device, which is a new version of the Guided Growth Plate System (GGPS) from which it differs for small modifications compared to the original design. The purpose of the study is to collect clinical evidence from the use of the device in a representative number of pediatric patients who have already been treated with the device in the study and with at least one control visit post removal of plaque..

For this purpose, a retrospective PMCF study was considered to be the most appropriate study design to obtain the necessary information.

DETAILED DESCRIPTION:
Guided Growth Plate System Plus (also named 8 Plate Plus) has been developed to redirect long bone growth and is used to correct gradually angular deformity in growing children. The device is indicated for the treatment of specific conditions/pathologies between which:

* deformity of the knee (femur and / or tibia) in varum/valgus or flexural extension;
* deformity of the ankle in varum/valgus or plantar flexion;
* femur and/or tibia length discrepancy.

Objectives:

The primary objective of the clinical investigation is to assess the safety of the 8 Plate Plus.

The secondary objective of the clinical investigation is to assess the clinical benefit of the 8 Plate Plus.

The Investigator will include in the study the patients who at the screening visit (Visit 0) will meet all the selection criteria. It is understood that, given the retrospective nature of the study and given that the consent of eligible patients has been collected in advance, the patient should not attend the screening visit or subsequent visits. In addition, during the screening visit (Visit 0) the Investigator will collect demographic data and patient history.

Subsequently, the data of interest relating to the surgery for the application of the plate (Visit 1) and the period of treatment will be collected, or related to the 2 follow up visits (Visits 2 and 3) carried out until or at the removal of the plate/ plates (Visit 4).

The course of treatment will be monitored as per clinical practice and will then be collected data that correspond to the follow-up visit planned on average 4 months after removal of the plate/plates (visit 5).

ELIGIBILITY:
Inclusion Criteria:

* he/she has been diagnosed with an angular deformity or discrepancy in length of femur and/or tibia
* at the time of treatment he/she had not yet reached the age of 18;
* at the time of treatment the growth plates of the treated limbs was not already closed;
* according to the Investigator's judgment, angular deformity and/or length discrepancy had a regular indication for surgical treatment with tensioning plates
* deformity was treated with the 8 Plate Plus , according to the manufacturer's instructions
* the treatment with 8 Plate Plus was completed and the patient had at least one post-removal control of the plate
* clinical patient data for the evaluation of safety and benefit of the device are still available

Exclusion Criteria:

* Not treated with 8 Plate Plus to correct upper limb deformities only and not lower limb deformities
* its clinical data are no longer accessible and /or do not allow the evaluation of the safety and benefit of the device under study
* had a medical condition which constitutes a contraindication to treatment with 8 Plate Plus in accordance with the manufacturer's instructions for use;
* at the same time was treated with an unauthorised device which could not be removed without putting the patient's safety at risk.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Paediatric patients with open physis (growing children) who have been diagnosed with an angular deformity or discrepancy in length of femur and/or tibia.
  Patients must not be over 18 years of age at the time of implantation.
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pediatric patients treated with Guided Growth Plate System Plus
Started | 69
Completed | 69
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pediatric Patients Treated With Guided Growth Plate System Plus
Number analyzed (Participants) | 69
Age, Customized [Mean (Standard Deviation); unit: years]
  Age of partecipants | 11.9 (1.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 69
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 69

OUTCOME MEASURES:

1. Primary Outcome: Safety Measurement: Percentage of Subjects Who During the Observation Period Have at Least One Complication Certainly or Potentially Related to the Device in the Studio
Description: Such complications shall be understood as:
  * a serious adverse event expected or not expected
  * a hardware failure (for example, breaking, detaching or folding of the plate or screws).
Time Frame: an average of 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Pediatric patients treated with Guided Growth Plate System Plus: Non-skeletally mature children with deformities of the long bones of the lower limbs.
Arm/Group | Pediatric patients treated with Guided Growth Plate System Plus
Number analyzed (Participants) | 69
Participants | 12

2. Secondary Outcome: Efficacy Measurement: the Percentage of Subjects That During the Observation Period Have Achieved the Treatment Objectives
Description: The treatment objectives are defined as:
  * for hemiepiphysiodesis, partially or completely corrected angular deformity of the femur and/or tibia in the direction of standard alignment (normal values of mMPTA and mLDFA between 85° and 89°);
  * for epiphysiodesis, discrepancy in the length of the femur and/or tibia partially or completely corrected with respect to the morphologically normal length of the contralateral limb.
Time Frame: an average of 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric patients treated with Guided Growth Plate System Plus
Number analyzed (Participants) | 69
Participants | 68

ADVERSE EVENTS:
Time Frame: from the application of the plate to first post-removal visit: 2 years
Arm/Group | Pediatric patients treated with Guided Growth Plate System Plus
All-Cause Mortality (participants affected / at risk) | 0/69
Serious Adverse Events (participants affected / at risk) | 0/69
Other Adverse Events (participants affected / at risk) | 12/69
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pediatric patients treated with Guided Growth Plate System Plus (N=69)
hypertrophic scar (Skin and subcutaneous tissue disorders) | 2 (2)
mild medial swelling (Skin and subcutaneous tissue disorders) | 1 (1)
Superficial infection (Infections and infestations) | 1 (1)
slight limitation of knee extension (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
wound bleeding (Vascular disorders) | 1 (1)
Stiffness (Musculoskeletal and connective tissue disorders) | 2 (2)
keloid scarring (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/91/NCT05241691/Prot_SAP_000.pdf